CLINICAL TRIAL: NCT01175629
Title: CSP #569 - A Twin Study of the Course and Consequences of PTSD in Vietnam Era Veterans
Brief Title: Veteran Health Study
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 569
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Stress Disorders, Post-Traumatic; Depression; Diabetes; Cardiovascular Disease
Keywords: Stress Disorders, Post-Traumatic; Depression; Diabetes; Cardiovascular Disease; Depressive Disorder; Behavioral Symptoms; Metabolic Diseases; Mental Disorders; Anxiety Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Diabetes Mellitus; Cardiovascular Diseases; Depressive Disorder; Behavioral Symptoms; Metabolic Diseases; Mental Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: The Vietnam Era Twin (VET) Registry is a closed cohort composed of 7,369 middle-aged male-male twin pairs both of whom served in the military during the time of the Vietnam conflict (1965-1975). The Registry is a United States Department of Veterans Affairs resource that was originally constructed from military records; the Registry has been in existence for more than 15 years. It is one of the largest national twin registries in the US and currently has subjects living in all 50 states. Initially formed to address questions about the long-term health effects of service in Vietnam the Registry has evolved into a resource for genetic epidemiological studies of mental and physical health conditions. Several waves of mail and telephone surveys have collected a wealth of health-related information on Registry twins. Other data collection efforts have focused on specific sets of twin pairs and conducted detailed clinical or laboratory testing.

SUMMARY:
The purpose of The Veteran Health Study (CSP #569) is to better understand the mental and physical health of veterans as they get older. We are inviting approximately 10,000 members of the Vietnam Era Twin (VET) Registry to participate. As veterans approach their mid-sixties, it is important to understand the impact of wartime deployment on health and mental health outcomes nearly 40 years later.

The investigators will assess the prevalence of post-traumatic stress disorder (PTSD) and other mental and physical health conditions for Vietnam era veterans, and explore the relationship between PTSD and other conditions.

CSP #569 involves 3 phases of data collection. In Phase I, VET Registry members are invited to complete a paper and pencil questionnaire including items on physical and mental health, disability, health behaviors, demographic information and use of health care services. After completing Phase I, VET Registry members are invited to Phase II which involves a telephone interview about mental health. In Phase III, some of those who participated in Phase I will be invited to a sub-study confirming self-reported heart disease and diabetes using a provider survey.

Data collected for CSP #569 will be combined with existing VET Registry data. This will provide a rich picture of the health of Vietnam era veterans and the influence of PTSD on the lives of veterans.

ELIGIBILITY:
Inclusion Criteria:

* All twins who are currently active in the VET Registry will be invited to participate in CSP #569.

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects are members of the Vietnam Era Twin Registry, and are males born between 1939-1957.
Sampling Method: Non-Probability Sample
Enrollment: 7568 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of lifetime and current psychiatric conditions including PTSD in Vietnam Era Twin Registry members who served during the Vietnam Era. | two years

SECONDARY OUTCOMES:
Characterize the physical health of Vietnam Era Twin Registry members who served during the Vietnam Era. | two years
Characterize the level of current disability in Vietnam Era Twin Registry members who served during the Vietnam Era. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jack H Goldberg, PhD MA BA, Study Chair — VA Puget Sound Health Care System, Seattle; Kathryn M. Magruder, PhD MPH BA, Study Chair — Ralph H Johnson VA Medical Center, Charleston
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Result] Magruder K, Yeager D, Goldberg J, Forsberg C, Litz B, Vaccarino V, Friedman M, Gleason T, Huang G, Smith N. Diagnostic performance of the PTSD checklist and the Vietnam Era Twin Registry PTSD scale. Epidemiol Psychiatr Sci. 2015 Oct;24(5):415-22. doi: 10.1017/S2045796014000365. Epub 2014 Jun 6. PMID 24905737
- [Result] Vaccarino V, Goldberg J, Magruder KM, Forsberg CW, Friedman MJ, Litz BT, Heagerty PJ, Huang GD, Gleason TC, Smith NL. Posttraumatic stress disorder and incidence of type-2 diabetes: a prospective twin study. J Psychiatr Res. 2014 Sep;56:158-64. doi: 10.1016/j.jpsychires.2014.05.019. Epub 2014 Jun 9. PMID 24950602
- [Result] Goldberg J, Magruder KM, Forsberg CW, Kazis LE, Ustun TB, Friedman MJ, Litz BT, Vaccarino V, Heagerty PJ, Gleason TC, Huang GD, Smith NL. The association of PTSD with physical and mental health functioning and disability (VA Cooperative Study #569: the course and consequences of posttraumatic stress disorder in Vietnam-era veteran twins). Qual Life Res. 2014 Jun;23(5):1579-91. doi: 10.1007/s11136-013-0585-4. Epub 2013 Dec 7. PMID 24318083